CLINICAL TRIAL: NCT01503229
Title: Open Label Pharmacodynamic Study of Abiraterone Acetate in the Treatment of Metastatic, Castration Resistant Prostate Cancer
Brief Title: Abiraterone Acetate in Treating Patients With Metastatic Hormone-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Bruce Montgomery, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7639; NCI-2011-03745 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0801; 7639 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); NCT01508234 (obsolete NCT alias)
Record Dates: First submitted 2011-12-27; First posted 2012-01-02 (Estimated); Results first posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: Hormone-Resistant Prostate Cancer; Metastatic Prostate Carcinoma; Recurrent Prostate Carcinoma; Stage IV Prostate Adenocarcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone; deltacortene; prednylidene

ARMS (1):
- Treatment (abiraterone acetate and prednisone) (Experimental): Patients receive abiraterone acetate orally once daily and prednisone orally twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Abiraterone Acetate; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone Acetate — Given by mouth
  Other Names: CB7630; Zytiga
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone; SK-Prednisone

SUMMARY:
This phase II trial studies how well abiraterone acetate works in treating patients with hormone-resistant prostate cancer that has spread from the primary site (place where it started) to other places in the body (metastatic). Abiraterone acetate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the magnitude of tissue testosterone suppression by abiraterone acetate in metastatic castrate-resistant prostate cancer (CRPC) (resistant to luteinizing hormone-releasing hormone [LHRH] agonist or orchiectomy ± antiandrogen) after one month of treatment to establish tissue based mechanism of action.

OUTLINE:

Patients receive abiraterone acetate orally once daily and prednisone twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Have signed an informed consent document indicating that the subjects understands the purpose of and procedures required for the study and are willing to participate in the study
* Written authorization for use and release of health and research study information has been obtained
* Be willing/able to adhere to the prohibitions and restrictions specified in this protocol
* Able to swallow the study drug whole as a tablet
* Willing to take abiraterone acetate on an empty stomach; no food should be consumed at least two hours before and for at least one hour after the dose of abiraterone acetate is taken
* Patients who have partners of childbearing potential must be willing to use a method of birth control with adequate barrier protection as determined to be acceptable by the principal investigator and sponsor during the study and for 1 week after last dose of abiraterone acetate
* Histologically proven adenocarcinoma of the prostate
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Metastatic castration resistant prostate cancer as defined by serum testosterone < 50 ng/ml and one of the following:

  * Prostate specific antigen (PSA) level of at least 2 ng/ml that has risen on at least 2 successive occasions at least 1 week apart
  * Evaluable disease progression by modified RECIST (Response Evaluation Criteria in Solid Tumors)
  * Progression of metastatic bone disease on bone scan with > 2 new lesions
* Maintenance of Lupron or antagonist unless previously treated with orchiectomy
* The presence of metastatic disease amenable to computed tomography (CT) or ultrasound guided biopsy; this may include thoracolumbar vertebral bodies, pelvis, femur or humerus, or soft tissue or nodal metastasis amenable to biopsy (excluding lung or pleural lesions)
* Patients may have received secondary hormonal manipulations (excluding prior abiraterone acetate, MDV3100 or TAK700) or up to two lines of chemotherapy; all prior therapy except Lupron must have been discontinued for more than 4 weeks before enrollment
* Serum potassium of >= 3.5 mEq/L
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) < 1.5 x upper limit of normal (ULN)
* Bilirubin levels < 1.5 x ULN
* Serum albumin of >= 3.0 g/dL
* Total bilirubin =< 1.5 x ULN
* Calculated creatinine clearance >= 60 mL/min
* Platelet count of >= 100,000/uL
* Absolute neutrophil count of > 1,500 cell/mm^3
* Hemoglobin >= 9.0 g/dL

Exclusion Criteria:

* Active infection or other medical condition that would make prednisone/prednisolone (corticosteroid) use contraindicated
* Patients who are currently receiving active therapy for other neoplastic disorders will not be eligible
* Patients with histologic evidence of small cell carcinoma of the prostate will not be eligible
* Known brain metastasis
* Uncontrolled hypertension (systolic blood pressure [BP] >= 160 mmHg or diastolic BP >= 95 mmHg); patients with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive treatment
* Active or symptomatic viral hepatitis or chronic liver disease
* History of pituitary or adrenal dysfunction
* Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) class II-IV heart disease or cardiac ejection fraction measurement of < 50 % at baseline
* Atrial fibrillation, or other cardiac arrhythmia requiring medical therapy
* Administration of an investigational therapeutic within 30 days of screening
* Patients with dementia/psychiatric illness/social situations that would limit compliance with study requirements or would prohibit the understanding and/or giving of informed consent will not be eligible
* Patients with any condition that, in the opinion of the investigator, would compromise the well-being of the subject or the study or prevent the subject from meeting or performing study requirements
* Patients requiring therapeutic anticoagulation (e.g., warfarin, dabigatran, heparin, or low molecular weight heparins [Lovenox, dalteparin])
* Patients with poorly controlled diabetes
* Patients with a history of gastrointestinal disorders (medical disorders or extensive surgery) that may interfere with the absorption of the study agents
* Patients with a pre-existing condition that warrants long-term corticosteroid use in excess of study dose
* Patients with known allergies, hypersensitivity, or intolerance to abiraterone acetate or prednisone or their excipients
* Child-Pugh class B or C hepatic impairment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Montgomery, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Abiraterone Acetate and Prednisone): Patients receive abiraterone acetate daily and prednisone twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Abiraterone Acetate: Given orally
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
  Prednisone: Given orally
Period: Overall Study
Arm/Group | Treatment (Abiraterone Acetate and Prednisone)
Started | 30
Completed | 29
Not Completed | 1
Not completed — Withdrew consent | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Abiraterone Acetate and Prednisone)
Number analyzed (Participants) | 29
Age, Customized [Median (Full Range); unit: years]
  Age of participants | 71 [44 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 25
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Change in Tissue Testosterone and Dihydrotestosterone
Description: Tissue testosterone will be measured in biopsy tissues
Time Frame: From baseline to week 4
Measure: Median (95% Confidence Interval); unit: pg/mg
Arm/Group | Treatment (Abiraterone Acetate and Prednisone)
Number analyzed (Participants) | 29
pg/mg | 0.156 [0.019 to 0.168]

ADVERSE EVENTS:
Time Frame: Serious adverse events only were collected over the duration of the study from enrollment through disenrollment for the last patient. Total maximum time on study was 2 years.
Description: No adverse events beyond SAE were collected given that the medication was standard of care. SAE were tracked related to any morbidity related to biopsy
Groups:
- Treatment (Abiraterone Acetate and Prednisone): Patients receive abiraterone acetate orally once daily and prednisone orally twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Abiraterone Acetate: Given by mouth
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
  Prednisone: Given by mouth
Arm/Group | Treatment (Abiraterone Acetate and Prednisone)
All-Cause Mortality (participants affected / at risk) | 29/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT01503229/Prot_SAP_000.pdf